CLINICAL TRIAL: NCT03448757
Title: Determination of Autonomic Responses to the Exposure of Low Energy Electromagnetic Fields With Frequency Modulation in Patients With Advanced Hepatocellular Carcinoma and Healthy Individuals.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Frederico Perego Costa, Principal investigator, Hospital Sirio-Libanes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSL 2016-83
Record Dates: First submitted 2018-02-20; First posted 2018-02-28 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: LEEF; hemodynamic parameters; heart beat; biofeedback effect
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: measuring hemodynamic parameters heart beat to heart beat during single-frequency exposure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autonomic response (Experimental): Group for determination of biofeedback response - 40 individuals. For the formation of this study group of subjects, 20 healthy volunteers and 20 patients with advanced hepatocellular carcinoma will be selected and studied.
  Group for determination of ideal frequency - 20 patients. For the formation of this study group of subjects, 20 patients with advanced hepatocellular carcinoma participants in the group will be selected and studied to determine biofeedback response.
  Group for determination of new specific frequencies - 20 individuals. For the formation of this study group of subjects, 20 patients with advanced hepatocellular carcinoma not exposed to any specific frequency will be selected.
  Interventions: Other: measuring hemodynamic parameters heart beat to heart beat during single-frequency exposure

INTERVENTIONS:
Other: measuring hemodynamic parameters heart beat to heart beat during single-frequency exposure — This study aims to create a method for non-invasive diagnosis of biofeedback effect exposure to LEEF modulated to specific frequencies in individuals exposed to hepatocellular carcinoma -specific frequencies in increasing sequential manner, frequency to frequency in patients with advanced hepatocellular carcinoma and healthy individuals.
  Patients with advanced hepatocellular carcinoma will be exposed to specific LEEF-modulated frequencies (3 to 10 Hz difference) to identify the optimal frequency associated with greater response to the biofeedback effect in patients with advanced hepatocellular carcinoma.

SUMMARY:
Biofeedback is an autonomic response observed during the exposure period to CEMBE. After prospectively evaluating 20 healthy individuals or 40 patients with advanced breast cancer or hepatocarcinoma, it was possible to determine subtle hemodynamic changes consistent with the biofeedback effect associated with exposure to a cancer-specific set of modulated frequencies.

Once CEMBE is administered through an intra-oral administration device, the human body absorbs the energy applied at the level of 0.2-1 mW / kg, with a peak absorption in 10 g of tissue between 55 and 132 mW / kg. Initially, the discriminatory study analyzing 9 hemodynamic parameters recorded beat heart beat in 18 individuals demonstrated a hemodynamic pattern specific for hepatocarcinoma and breast cancer, with sensitivity of 94.1% and 95%, respectively, and specificity of 75% and 95%, respectively. These findings were validated in blind analysis in the remaining 56 patients, confirming the high rate of discriminatory success.

A specific pattern of response associated with exposure of a cancer-specific frequency group was also observed in patients diagnosed with neoplasia, since the control group of healthy individuals did not present these response patterns.

This specific signature of response to CEMBE-modulated exposure to cancer-specific frequencies was significantly altered only in patients with hepatocarcinoma after tumor withdrawal (Costa et al, 2015a).

DETAILED DESCRIPTION:
This is an exploratory, national, unicentric, open study, to be conducted at the Instituto de Ensino e Pesquisa do Hospital Sírio Libanês, aiming to determine a method of prospective measurement of autonomic responses resulting from exposure to LEEF modulated at specific frequencies and with sequential exposure (frequency to frequency) in healthy individuals and patients with advanced hepatocellular carcinoma , followed by new exposure with a new set of specific frequencies determined by mathematical method.

This study aims to create a method for non-invasive diagnosis of biofeedback effect exposure to LEEF modulated to specific frequencies in individuals exposed to hepatocellular carcinoma -specific frequencies in increasing sequential manner, frequency to frequency in patients with advanced hepatocellular carcinoma and healthy individuals.

Patients with advanced hepatocellular carcinoma will be exposed to specific LEEF-modulated frequencies (3 to 10 Hz difference) to identify the optimal frequency associated with greater response to the biofeedback effect in patients with advanced hepatocellular carcinoma.

Patients with advanced hepatocellular carcinoma will be exposed to modulated LEEF at a new set of specific frequencies determined by mathematical method to identify biofeedback effect in patients with advanced hepatocellular carcinoma.

This study does not propose to study a therapeutic procedure. For this reason, no evolutionary clinical data will be analyzed during and after study intervention.

This study will be conducted in an outpatient setting and is expected to last 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

  * Must be considered healthy, with no known relevant comorbidity.
  * Patients must not be carriers of active malignant neoplasm or have a history of malignant neoplasm.
  * Must be over 18 years old.
  * Must have the ability to understand and provide written Informed Consent.

Patients with hepatocellular carcinoma

* Patients must be diagnosed with inoperable HCC.
* Presence of the primary or metastatic tumor at the time of the procedure.
* Patients diagnosed with hepatic cirrhosis must be restricted to Child-Pugh A or B.
* Patients with AFP> 400 ng/ml and characteristic image do not need histopathological confirmation. However, in patients with serology for active B virus, this AFP value must be greater than 4000 ng/ml. The remaining patients must have histological confirmation of HCC.
* Patients may be in observation or in the course of systemic or intra-hepatic treatment.
* Must have the ability to understand and provide written Informed Consent.

Exclusion Criteria:

* Individuals selected for this study will be excluded if they meet the following exclusion criteria:

  * They cannot stop antihypertensive drugs or beta blockers for at least 24 hours.
  * Have a pacemaker or other implantable device.
  * Pregnant or breastfeeding.
  * Under the age of 18.
  * Patients undergoing radiotherapy or up to 2 weeks after its suspension.
  * Inability to understand and provide written Informed Consent.
  * Child Pugh C hepatic cirrhosis.
  * Patient without definite diagnosis.
  * Absence of primary or metastatic tumor at the time of the procedure.

Potentially eligible participants will be previously guided by the researcher on the objectives and risks of the study in question and will be presented and informed about the Free, Prior and Informed Consent document.

Only after all doubts related to the study have been clarified and the Free, Prior and Informed Consent document has been signed, will the study participant be invited and scheduled to attend the Oncology Center clinic of Hospital Sírio Libanês.

Patients must be informed that they may not drink alcohol up to 12 hours before the procedure, as there may be interference during the procedure.

They will also be advised not to use antihypertensive drugs like beta-blockers or calcium channel inhibitors 24 hours before the procedure, without resulting in a risk to the participant's health.

In this study, following or follow-up of patients is not foreseen.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2023-12-16 (Estimated)

PRIMARY OUTCOMES:
non-invasive hemodynamic parameter measurements during exposure AM RF EMF | 90 min on day 1 and day 2
  Identification of hemodymanic alterations induced by the exposure to low levels of amplitude modulation radiofrequency electromagnetic fields (AM RF EMF) in healthy individuals and patients with advanced hepatocellular carcinoma using Artificial Intelligence program to analyze the recorded data set collected by a high-precision and non-invasive hemodynamic monitor.

SECONDARY OUTCOMES:
Hemodynamic alteration´s comparison among advanced cancer patients and healthy controls | 120 min (single procedure)
  Comparison of hemodynamic alteration during exposure to a group of hepatocellular-specific AM RF EMF recorded in healthy individuals and patients with advanced hepatocellular carcinoma using Artificial Intelligence algorithms to compare the recorded data set collected by a high-precision and non-invasive hemodynamic monitor.

OTHER OUTCOMES:
Searching for cancer-specific frequency modulation | 120 min (single procedure)
  Identification of specifc hemodynamic alteration recorded during the exposure to a series of specific frequency modulations AM RF EMF recorded in healthy individuals and patients with advanced hepatocellular carcinoma using Artificial Intelligence program.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Sírio-Libanês, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no sharing plan.